CLINICAL TRIAL: NCT04309682
Title: Clinical and Radiographic Evaluation of Implants Placed Without Bone Grafts in Two Different Sinus Floor Elevation Techniques. A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Implants Placed Without Bone Grafts in Two Different Sinus Floor Elevation Techniques.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Clinical Director of Implant Program - Periodontology and Implantology Consultant, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PER8273004
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Dental Implant Placement
Keywords: Crestal sinus approach; lateral sinus approach; implant stability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- crestal sinus approach technique (Experimental): Full thickness flap will be elevated at the edentulous site with two vertical releasing incision and then the preparation of osteotomy will be prepared following standard implant system protocol preparation of the osteotomy. Drilling will be done gently till reaching 0-1mm from the sinus floor, then implant placement will take place and the implant itself will be used to gently elevate the sinus up to 3-5mm
  Interventions: Procedure: crestal sinus approach technique
- lateral sinus elevation technique (Active Comparator): a full-thickness flap will be elevated at the edentulous site with two vertical releasing incisions extending to the vestibule for better reflection and exposure to the lateral wall of the sinus. The lateral antrostomy will be prepared in the lateral sinus wall using rotary bur no. 8 to provide adequate access to remove the thin to thick cortical bone and to expose the thin sinus membrane. The membrane will be elevated across the sinus floor and up the medial wall and this elevation must extend anteriorly-posteriorly to provide the exposed sinus floor. Drilling will be done gently till reaching 0-1mm from the sinus floor, then implant placement will take plac
  Interventions: Procedure: Lateral sinus approach

INTERVENTIONS:
Procedure: crestal sinus approach technique — a Full thickness flap will be elevated at the edentulous site with two vertical releasing incision and then the preparation of osteotomy will be prepared following standard implant system protocol preparation of the osteotomy. Drilling will be done gently till reaching 0-1mm from the sinus floor, then implant placement will take place and the implant itself will be used to gently elevate the sinus up to 3-5mm.
  Other Names: zimmer biomed dental implants and crestal sinus approach
  Arms: crestal sinus approach technique
Procedure: Lateral sinus approach — a full-thickness flap will be elevated at the edentulous site with two vertical releasing incisions extending to the vestibule for better reflection and exposure to the lateral wall of the sinus. The lateral antrostomy will be prepared in the lateral sinus wall using rotary bur no. 8 to provide adequate access to remove the thin to thick cortical bone and to expose the thin sinus membrane. The membrane will be elevated across the sinus floor and up the medial wall and this elevation must extend anteriorly-posteriorly to provide the exposed sinus floor. Drilling will be done gently till reaching 0-1mm from the sinus floor, then implant placement will take place
  Other Names: Zimmer biomed dental implants and lateral sinus approach
  Arms: lateral sinus elevation technique

SUMMARY:
Statement of the problem: Vertical bone height reduction after extraction in the posterior maxilla complicates the treatment plan. Lateral sinus elevation, crestal sinus elevation, using short implants and different grafting procedures are some of the proposed treatment protocols, however, there is still a gap of knowledge in high quality evidence for the most effective approach. Purpose : The aim of the study is to evaluate clinical long term implant stability and radiographic vertical bone height gain after implant placement in posterior maxilla using crestal sinus approach in comparison to lateral sinus elevation technique. Materials and Methods: Thirty patients have single maxillary posterior tooth in atrophic maxilla will be enrolled. Patients will be allocated randomly into two groups; group 1 (test group) will receive implants using crestal sinus approach and group 2 (control group) will be assigned to the lateral sinus elevation technique, no bone grafts will be placed in both groups. Resonance frequency analysis will be employed to measure implant stability with a dedicated device (Osstell). For each implant, implant stability quotient ISQ values will be measured from the four sites.The mean of all measurements will be rounded to a whole number and regarded as the final ISQ of the implant. ISQ values will be obtained after implant insertion, at 3 months after delivery of the final restoration, at 6 and 12 months post-surgical. CBCT will be taken at 3 &12 months follow up periods, to assess the amount of bone height gained around the dental implants in both groups.

DETAILED DESCRIPTION:
1. Clinical examination and preoperative evaluation using CBCT:

   1. Evaluation of the patient's general condition of the oral cavity, to make sure it complies with the criteria required to be enrolled in the study in terms of oral hygiene, pathological conditions, occlusion and inter-arch space.
   2. A preoperative CBCT will be performed for each patient prior to the surgery. Evaluation of available bone height and bucco-palatal bone width. Suitable implant length and diameter will be determined as well.
2. Random allocation: The patients will be divided into two groups with random allocation. Allocation ratio is 1:1. Randomization list will be provided using computerized excel sheet and will be concealed to the principle investigator till the time of the surgery, and will be kept with a contributor (Ingy Kastour) a clinician in IDCE who is not involved in the trial procedures. A phone call will be done after administration of anesthesia to reveal the randomization sequence for each case.
3. Blinding: The outcome assessors will be blinded, the outcome assessor (CoI-II) for the implant stability and the outcome assessor (CoI-V) for the vertical bone height difference obtained from blinded CBCTs, outcome assessor (CoI-III) of the other variables will be also blinded. Blinding of the principle investigator and participants cannot be achieved due to different surgical procedures
4. Surgical procedure:

   After administration of local anesthesia, the allocation will be revealed, for the test group, a Full thickness flap will be elevated at the edentulous site with two vertical releasing incision and then the preparation of osteotomy will be prepared following standard implant system protocol preparation of the osteotomy. Drilling will be done gently till reaching 0-1mm from the sinus floor, then implant placement will take place and the implant itself will be used to gently elevate the sinus up to 3-5mm. For the control group, a full-thickness flap will be elevated at the edentulous site with two vertical releasing incisions extending to the vestibule for better reflection and exposure to the lateral wall of the sinus. The lateral antrostomy will be prepared in the lateral sinus wall using rotary bur no. 8 to provide adequate access to remove the thin to thick cortical bone and to expose the thin sinus membrane. The membrane will be elevated across the sinus floor and up the medial wall and this elevation must extend anteriorly-posteriorly to provide the exposed sinus floor. Drilling will be done gently till reaching 0-1mm from the sinus floor, then implant placement will take place. Primary stability of the implant will be measured by rotational insertion torque value, to be ≥30Ncm(25). A resorbable collagen membrane will be placed over the window preparation in the lateral approach to prevent the flap tissue in cooperating inside the antrostomy and the osseointegration process. Primary closure of the flap will be achieved.
5. Postoperative Care:

   1. Antibiotics (Amoxicillin 1g orally- twice daily for 5 days).
   2. Anti-inflammatory drugs (NSAIDS; Ibuprofen 600mg three times daily for 5 days).
   3. Antiseptic mouth rinse (0.12% Chlorhexidine oral rinse) will be prescribed starting from the second day for 60 seconds, 15 ml each time, two times a day for 14 days.
   4. Patient self-care instructions:

      * Application of an ice bag to the treated area for the first 24 hours will be instructed.
      * The patients will be instructed to gently brush the operated area after two weeks with a soft brush.
      * In case of emergency; severe pain and bleeding, the patient will call the co-investigator and will be presented to the clinic.
      * Patients will be recalled after two weeks for suture removal and every month for supportive periodontal therapy and recording of outcome variables at three, six and twelve months.

After 3 months of the implant placement, stage II will be performed, 2 weeks later, impressions will be taken as regular for the prosthetic crowns fabrication. All crowns will be temporary cemented to allow an easy access to the implant platform for the follow-up RFA measurements.

ELIGIBILITY:
Inclusion Criteria:

1 Patients who have at least one missing posterior maxillary tooth. 2. Adults above the age of 18. 3. Bone height from 4mm to 6mm under the maxillary sinus assessed in CBCT. 4. Good oral hygiene. 5. Patient accepts to sign an informed consent.

Exclusion Criteria:

1. Smokers.
2. Pregnant and lactating females
3. Medically compromised patients. as Uncontrolled diabetic patients, patients taking bisphosphonates injection for treatment of osteoporosis, patients with active cardiac diseases, patients undergoing radiotherapy or chemotherapy, or any other medical and general contraindications for the surgical procedure (i.e. ASA score ≥III)
4. Patients with active infection related at the site of implant/bone graft placement.
5. Patients with untreated active periodontal diseases.
6. Patients with parafunctional habits.
7. Acute or chronic sinusitis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Long term Implant stability | 3 - 6 - 12 months
  Implant stability will be measured using Osstell to assess any changes in the implant stability over time and changes from baseline

SECONDARY OUTCOMES:
Vertical bone height gain | 3 - 12 months
  Measured by CBCT
Post-surgical pain | for 10 days after the surgery
  Measured using Visual Analogue Scale (VAS) The patients will mark the pain perception in a non-numerical 100 mm line ranging from "no pain=0" (left) to "very painful=100" (right).
Patient satisfaction regarding the function | 12 months
  Measured using Visual Analogue Scale (VAS) The patients will mark their satisfaction in a non-numerical 100 mm line ranging from "not at all satisfied=0" (left) to "very satisfied=100" (right), for each implant.
Plaque Index | 3 - 6 - 12 months
  Periodontal probe
Modified Bleeding Index | 3 - 6 - 12 months
  Periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed I Abo El Futtouh, Master, Principal Investigator — Clinical Director of Implant Program - Misr International University; Inas M El-Zayat, Doctor, Study Director — Assoc. Professor - Operative department, Misr International University; Mariam S Hanna, Bsc, Study Director — Dentist/Researcher - IDCE; Nael A Mina, Bsc, Study Chair — Misr International University; Abdel Rahman A Abdel Rahman, Master, Study Chair — International Dental Contiuing Education
Locations (1):
- International Dental Continuing Education (IDCE) centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data can be shared
Supporting Information: SAP, CSR
Time Frame: One year
Access Criteria: Principal investigator

REFERENCES:
- [Background] ROSEN MD, SARNAT BG. Change of volume of the maxillary sinus of the dog after extraction of adjacent teeth. Oral Surg Oral Med Oral Pathol. 1955 Apr;8(4):420-9. doi: 10.1016/0030-4220(55)90111-0. No abstract available. PMID 14370769
- [Background] Sharan A, Madjar D. Maxillary sinus pneumatization following extractions: a radiographic study. Int J Oral Maxillofac Implants. 2008 Jan-Feb;23(1):48-56. PMID 18416412
- [Background] Misch CE, Steignga J, Barboza E, Misch-Dietsh F, Cianciola LJ, Kazor C. Short dental implants in posterior partial edentulism: a multicenter retrospective 6-year case series study. J Periodontol. 2006 Aug;77(8):1340-7. doi: 10.1902/jop.2006.050402. PMID 16937587
- [Background] de Sa e Frias V, Toothaker R, Wright RF. Shortened dental arch: a review of current treatment concepts. J Prosthodont. 2004 Jun;13(2):104-10. doi: 10.1111/j.1532-849X.2004.04016.x. PMID 15210006
- [Background] Tatum H Jr. Maxillary and sinus implant reconstructions. Dent Clin North Am. 1986 Apr;30(2):207-29. PMID 3516738
- [Background] Boyne PJ, James RA. Grafting of the maxillary sinus floor with autogenous marrow and bone. J Oral Surg. 1980 Aug;38(8):613-6. No abstract available. PMID 6993637
- [Background] Zitzmann NU, Scharer P. Sinus elevation procedures in the resorbed posterior maxilla. Comparison of the crestal and lateral approaches. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Jan;85(1):8-17. doi: 10.1016/s1079-2104(98)90391-2. PMID 9474608
- [Background] Smiler DG. The sinus lift graft: basic technique and variations. Pract Periodontics Aesthet Dent. 1997 Oct;9(8):885-93; quiz 895. PMID 9573843
- [Background] Boyne PJ. Analysis of performance of root-form endosseous implants placed in the maxillary sinus. J Long Term Eff Med Implants. 1993;3(2):143-59. PMID 10146541
- [Background] Summers RB. A new concept in maxillary implant surgery: the osteotome technique. Compendium. 1994 Feb;15(2):152, 154-6, 158 passim; quiz 162. PMID 8055503
- [Background] Hallman M, Thor A. Bone substitutes and growth factors as an alternative/complement to autogenous bone for grafting in implant dentistry. Periodontol 2000. 2008;47:172-92. doi: 10.1111/j.1600-0757.2008.00251.x. No abstract available. PMID 18412581
- [Background] Marx RE, Carlson ER, Eichstaedt RM, Schimmele SR, Strauss JE, Georgeff KR. Platelet-rich plasma: Growth factor enhancement for bone grafts. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Jun;85(6):638-46. doi: 10.1016/s1079-2104(98)90029-4. PMID 9638695
- [Background] Lundgren S, Andersson S, Gualini F, Sennerby L. Bone reformation with sinus membrane elevation: a new surgical technique for maxillary sinus floor augmentation. Clin Implant Dent Relat Res. 2004;6(3):165-73. PMID 15726851
- [Background] Vercellotti T, De Paoli S, Nevins M. The piezoelectric bony window osteotomy and sinus membrane elevation: introduction of a new technique for simplification of the sinus augmentation procedure. Int J Periodontics Restorative Dent. 2001 Dec;21(6):561-7. PMID 11794567
- [Background] Srouji S, Kizhner T, Ben David D, Riminucci M, Bianco P, Livne E. The Schneiderian membrane contains osteoprogenitor cells: in vivo and in vitro study. Calcif Tissue Int. 2009 Feb;84(2):138-45. doi: 10.1007/s00223-008-9202-x. Epub 2008 Dec 9. PMID 19067018
- [Background] Jungner M, Legrell PE, Lundgren S. Follow-up study of implants with turned or oxidized surfaces placed after sinus augmentation. Int J Oral Maxillofac Implants. 2014 Nov-Dec;29(6):1380-7. doi: 10.11607/jomi.3629. PMID 25397801
- [Background] Aludden H, Mordenfeld A, Hallman M, Christensen AE, Starch-Jensen T. Osteotome-Mediated Sinus Floor Elevation With or Without a Grafting Material: A Systematic Review and Meta-analysis of Long-term Studies (>/=5-Years). Implant Dent. 2018 Aug;27(4):488-497. doi: 10.1097/ID.0000000000000798. PMID 30048350
- [Background] Ragab O, Fawzy El-Sayed KM, Zaki J, El-Khadem A, Shoeib M. Implant Survival in One-Stage Lateral versus Crestal Sinus Lift Procedures - A Systematic Review and Meta-Analysis. Indian J Sci Technol. 2017;10(13):1-10
- [Background] Bechara S, Kubilius R, Veronesi G, Pires JT, Shibli JA, Mangano FG. Short (6-mm) dental implants versus sinus floor elevation and placement of longer (>/=10-mm) dental implants: a randomized controlled trial with a 3-year follow-up. Clin Oral Implants Res. 2017 Sep;28(9):1097-1107. doi: 10.1111/clr.12923. Epub 2016 Jul 12. PMID 27402427
- [Background] Smeets EC, de Jong KJ, Abraham-Inpijn L. Detecting the medically compromised patient in dentistry by means of the medical risk-related history. A survey of 29,424 dental patients in The Netherlands. Prev Med. 1998 Jul-Aug;27(4):530-5. doi: 10.1006/pmed.1998.0285. PMID 9672946
- [Background] Chrcanovic BR, Kisch J, Albrektsson T, Wennerberg A. Factors Influencing Early Dental Implant Failures. J Dent Res. 2016 Aug;95(9):995-1002. doi: 10.1177/0022034516646098. Epub 2016 May 4. PMID 27146701
- [Background] Olmedo-Gaya MV, Manzano-Moreno FJ, Canaveral-Cavero E, de Dios Luna-del Castillo J, Vallecillo-Capilla M. Risk factors associated with early implant failure: A 5-year retrospective clinical study. J Prosthet Dent. 2016 Feb;115(2):150-5. doi: 10.1016/j.prosdent.2015.07.020. Epub 2015 Nov 3. PMID 26545864
- [Background] Vissink A, Spijkervet F, Raghoebar GM. The medically compromised patient: Are dental implants a feasible option? Oral Dis. 2018 Mar;24(1-2):253-260. doi: 10.1111/odi.12762. PMID 29480621
- [Background] Lobbezoo F, Brouwers JE, Cune MS, Naeije M. Dental implants in patients with bruxing habits. J Oral Rehabil. 2006 Feb;33(2):152-9. doi: 10.1111/j.1365-2842.2006.01542.x. PMID 16457676
- [Background] Testori T, Meltzer A, Del Fabbro M, Zuffetti F, Troiano M, Francetti L, Weinstein RL. Immediate occlusal loading of Osseotite implants in the lower edentulous jaw. A multicenter prospective study. Clin Oral Implants Res. 2004 Jun;15(3):278-84. doi: 10.1111/j.1600-0501.2004.01013.x. PMID 15142089
- [Background] Kim SH, Choi JH, Chung KR, Nelson G. Do sand blasted with large grit and acid etched surface treated mini-implants remain stationary under orthodontic forces? Angle Orthod. 2012 Mar;82(2):304-12. doi: 10.2319/032511-212.1. Epub 2011 Aug 10. PMID 21830933
- [Background] Koerich L, Weissheimer A, Koerich LE, Luz D, Deeb JG. A Technique of Cone-Beam Computerized Tomography Superimposition in Implant Dentistry. J Oral Implantol. 2018 Oct;44(5):365-369. doi: 10.1563/aaid-joi-D-17-00282. Epub 2018 May 2. No abstract available. PMID 29717909
- [Background] Cevidanes LH, Styner MA, Proffit WR. Image analysis and superimposition of 3-dimensional cone-beam computed tomography models. Am J Orthod Dentofacial Orthop. 2006 May;129(5):611-8. doi: 10.1016/j.ajodo.2005.12.008. PMID 16679201
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Background] Patil SP, Bhongade ML. Reviews of Complications from Lateral and Crestal Sinus Lifts Histologic Analysis. J Implant Adv Clin Dent. 2016;8